CLINICAL TRIAL: NCT02057575
Title: A Double-masked, Randomized, Controlled Study Assessing the Safety and Ocular Hypotensive Efficacy of PG324 Ophthalmic Solution, 0.01% and PG324 Ophthalmic Solution, 0.02%, Compared to AR-13324 Ophthalmic Solution, 0.02% and Latanoprost Ophthalmic Solution, 0.005% in Patients With Elevated Intraocular Pressure
Brief Title: Study Assessing Safety and Efficacy of PG324 Ophthalmic Solution in Patients With Elevated Intraocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG324-CS201
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Open Angle Glaucoma; Ocular Hypertension; Intraocular Pressure; AR13324; PG324
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — netarsudil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PG324 Ophthalmic Solution 0.01% (Experimental): Netarsudil 0.01%, Latanoprost 0.005% fixed combination ophthalmic solution
  Interventions: Drug: PG324 Ophthalmic Solution 0.01%
- PG324 Ophthalmic Solution 0.02% (Experimental): Netarsudil 0.02%, Latanoprost 0.005% fixed combination ophthalmic solution
  Interventions: Drug: PG324 Ophthalmic Solution 0.02%
- Netarsudil (AR-13324) Ophthalmic Solution 0.02% (Active Comparator): Netarsudil 0.02% ophthalmic solution
  Interventions: Drug: Netarsudil (AR-13324) Ophthalmic Solution 0.02%
- Latanoprost Ophthalmic Solution 0.005% (Active Comparator): Latanoprost 0.005% ophthalmic solution
  Interventions: Drug: Latanoprost Ophthalmic Solution 0.005%

INTERVENTIONS:
Drug: PG324 Ophthalmic Solution 0.01% — 1 drop in the evening (PM), once daily (QD), both eyes (OU)
  Arms: PG324 Ophthalmic Solution 0.01%
Drug: PG324 Ophthalmic Solution 0.02% — 1 drop in the evening (PM), once daily (QD), both eyes (OU)
  Arms: PG324 Ophthalmic Solution 0.02%
Drug: Netarsudil (AR-13324) Ophthalmic Solution 0.02% — 1 drop in the evening (PM), once daily (QD), both eyes (OU)
  Arms: Netarsudil (AR-13324) Ophthalmic Solution 0.02%
Drug: Latanoprost Ophthalmic Solution 0.005% — 1 drop in the evening (PM), once daily (QD), both eyes (OU)
  Arms: Latanoprost Ophthalmic Solution 0.005%

SUMMARY:
To evaluate the ocular hypotensive efficacy of PG324 ophthalmic solution relative to its individual components in patients with open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater.
* Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT)
* Corrected visual acuity in each eye equivalent to 20/200 or better
* Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

Ophthalmic:

* Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure, or narrow angles.
* Intraocular pressure >36 mmHg
* Known hypersensitivity to any component of the formulation, latanoprost, or to topical anesthetics.
* Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s)
* Refractive surgery in study eye(s)
* Ocular trauma within the six months prior to screening, or ocular surgery or laser treatment within the three months prior to screening.
* Evidence of ocular infection and inflammation
* Clinically significant ocular disease, which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe
* Central corneal thickness greater then 600 μm
* Any abnormality preventing reliable applanation tonometry of either eye

Systemic:

* Clinically significant abnormalities (as determined by the investigator) in laboratory tests at screening.
* Clinically significant systemic disease
* Participation in any investigational study within 30 days prior to screening
* Changes in systemic medication
* Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ramirez, M.S., Study Director — Aerie Pharmaceuticals, Inc.
Locations (23):
- United States (23):
  - Kenneth Sall, M.D., Artesia, California
  - United Medical Research Institute, Inglewood, California
  - Aesthetic Eye Care Institute, Newport Beach, California
  - Bacharach practice, Petaluma, California
  - Centre For Health Care, Poway, California
  - Clayton Eye Center, Morrow, Georgia
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Bradley Kwapiszeski, MD, Shawnee Mission, Kansas
  - Taustine Eye Center, Louisville, Kentucky
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Comprehensive Eye Care, St Louis, Missouri
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Rochester Ophthalmological Group, Rochester, New York
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Belmont, North Carolina
  - Michael E. Tepedino, M.D., High Point, North Carolina
  - The Eye Institute, Tulsa, Oklahoma
  - Texan Eye, Austin, Texas
  - Glaucoma Associates of Texas - Dallas Office, Dallas, Texas
  - Cataract & Glaucoma Center, El Paso, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Stacy R. Smith, M.D., Salt Lake City, Utah
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis RA, Levy B, Ramirez N, Kopczynski CC, Usner DW, Novack GD; PG324-CS201 Study Group. Fixed-dose combination of AR-13324 and latanoprost: a double-masked, 28-day, randomised, controlled study in patients with open-angle glaucoma or ocular hypertension. Br J Ophthalmol. 2016 Mar;100(3):339-44. doi: 10.1136/bjophthalmol-2015-306778. Epub 2015 Jul 24. PMID 26209587

RESULTS

PARTICIPANT FLOW:
Groups:
- PG324 Ophthalmic Solution 0.01%: PG324 Ophthalmic Solution 0.01%
  1 drop in the evening (PM), once daily (QD), both eyes (OU)
- PG324 Ophthalmic Solution 0.02%: PG324 Ophthalmic Solution 0.02%
  1 drop in the evening (PM), once daily (QD), both eyes (OU)
- Netarsudil (AR-13324) Ophthalmic Solution 0.02%: Netarsudil (AR-13324) Ophthalmic Solution 0.02%
  1 drop in the evening (PM), once daily (QD), both eyes (OU)
- Latanoprost Ophthalmic Solution 0.005%: Latanoprost Ophthalmic Solution 0.005%
  1 drop in the evening (PM), once daily (QD), both eyes (OU)
Period: Overall Study
Arm/Group | PG324 Ophthalmic Solution 0.01% | PG324 Ophthalmic Solution 0.02% | Netarsudil (AR-13324) Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Started | 74 | 73 | 78 | 73
Completed | 73 | 69 | 78 | 72
Not Completed | 1 | 4 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Dissallowed Concurrent Medication | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Latanoprost Ophthalmic Solution 0.005%: Latanoprost Ophthalmic Solution 0.005%
  1 drop daily in the evening (PM), once daily (QD), both eyes (OU)
- Total: Total of all reporting groups
Arm/Group | PG324 Ophthalmic Solution 0.01% | PG324 Ophthalmic Solution 0.02% | Netarsudil (AR-13324) Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005% | Total
Number analyzed (Participants) | 74 | 73 | 78 | 73 | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 35 | 33 | 28 | 125
  >=65 years | 45 | 38 | 45 | 45 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (11.26) | 64.2 (11.07) | 64.8 (11.28) | 65.1 (12.80) | 64.9 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 39 | 43 | 46 | 175
  Male | 27 | 34 | 35 | 27 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 20 | 15 | 14 | 64
  Not Hispanic or Latino | 59 | 53 | 63 | 59 | 234
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 3 | 1 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 10 | 17 | 12 | 54
  White | 56 | 62 | 58 | 60 | 236
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: The primary efficacy endpoint was the mean diurnal IOP across subjects within treatment group at Day 29.
Time Frame: Study treatment was administered for 28 days, and outcome measures collected on Day 29
Population: Modified intent to treat (mITT) population
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Netarsudil (AR-13324) Ophthalmic Solution: Netarsudil (AR-13324) Ophthalmic Solution
  1 drop in the evening (PM), once daily (QD), both eyes (OU)
- Latanoprost Ophthalmic Solution: Latanoprost Ophthalmic Solution
  1 drop in the evening (PM), once daily (QD), both eyes (OU)
Arm/Group | PG324 Ophthalmic Solution 0.01% | PG324 Ophthalmic Solution 0.02% | Netarsudil (AR-13324) Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 73 | 72 | 78 | 73
mmHg
  Day 1, Diurnal Mean | 25.11 (2.330) | 25.12 (2.374) | 25.35 (2.666) | 25.99 (2.828)
  Day 29, Diurnal Mean | 17.33 (2.770) | 16.52 (2.992) | 19.13 (3.219) | 18.44 (2.565)
Statistical Analysis 1: Comparison: PG324 Ophthalmic Solution 0.01% vs Netarsudil (AR-13324) Ophthalmic Solution; Test type: Superiority; p < 0.0001, t-test, 2 sided — PG324 0.01% vs netarsudil
Statistical Analysis 2: Comparison: PG324 Ophthalmic Solution 0.02% vs Netarsudil (AR-13324) Ophthalmic Solution; Test type: Superiority; p < 0.0001, t-test, 2 sided — PG324 0.02% vs. netarsudil
Statistical Analysis 3: Comparison: PG324 Ophthalmic Solution 0.01% vs Latanoprost Ophthalmic Solution; Test type: Superiority; p < 0.0001, t-test, 2 sided; PG324 0.01% vs. latanoprost
Statistical Analysis 4: Comparison: PG324 Ophthalmic Solution 0.02% vs Latanoprost Ophthalmic Solution; Test type: Superiority; p < 0.0001, t-test, 2 sided; PG324 0.02% vs. latanoprost

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected over the course of the study of the 28 day treatment period
Description: 1 Subject is not considered in the safety population; this subject was randomized but not treated. ( Number of subjects applies to All cause mortality, SAEs and other AEs sections)
Groups:
- Latanoprost Ophthalmic Solution: Latanoprost Ophthalmic Solution
  Latanoprost Ophthalmic Solution: 1 drop daily (evening)
Arm/Group | PG324 Ophthalmic Solution 0.01% | PG324 Ophthalmic Solution 0.02% | Netarsudil (AR-13324) Ophthalmic Solution | Latanoprost Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/73 | 0/78 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/73 | 0/78 | 3/73
Other Adverse Events (participants affected / at risk) | 46/73 | 55/73 | 49/78 | 12/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PG324 Ophthalmic Solution 0.01% (N=74) | PG324 Ophthalmic Solution 0.02% (N=73) | Netarsudil (AR-13324) Ophthalmic Solution (N=78) | Latanoprost Ophthalmic Solution (N=73)
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG324 Ophthalmic Solution 0.01% (N=73) | PG324 Ophthalmic Solution 0.02% (N=73) | Netarsudil (AR-13324) Ophthalmic Solution (N=78) | Latanoprost Ophthalmic Solution (N=73)
Conjunctival Hyperaemia (Eye disorders) | 29 (29) | 29 (29) | 27 (27) | 9 (9)
Lacrimation Increased (Eye disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Instillation Site Erythema (General disorders) | 11 (11) | 14 (14) | 17 (17) | 1 (1)
Instillation Site Pain (General disorders) | 5 (5) | 8 (8) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No